CLINICAL TRIAL: NCT04652869
Title: Mindfulness + tDCS to Reduce Urgency Incontinence in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia Conklin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Cynthia Conklin, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19110132; 1R21AG064361 (NIH)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Urinary Incontinence, Urge
Keywords: Transcranial Direct Current Stimulation (tDCS); Mindfulness; Situational Urge Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Transcranial Direct Current Stimulation; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Mindfulness Training (Experimental): Mindfulness training
  Interventions: Behavioral: Mindfulness
- Transcranial Direct Current Stimulation (tDCS) (Experimental): Transcranial direct current stimulation targeting the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation
- Mindfulness + tDCS (Experimental): Mindfulness training with transcranial direct current stimulation targeting the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation; Behavioral: Mindfulness

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation targeting the dorsolateral prefrontal cortex
  Other Names: tDCS
  Arms: Mindfulness + tDCS; Transcranial Direct Current Stimulation (tDCS)
Behavioral: Mindfulness — Mindfulness is a type of meditation in which you focus on being intensely aware of what you're sensing and feeling in the moment, without interpretation or judgment.
  Arms: Mindfulness + tDCS; Mindfulness Training

SUMMARY:
Urge urinary incontinence (UUI) is a common problem in older women, which vastly reduces quality of life. UUI sufferers frequently report situational triggers (e.g. approaching the front door) leading to urinary urgency and/or leakage, which can be caused by psychological conditioning. This project will test the feasibility, acceptability, and efficacy of brief mindfulness (MI) and non-invasive brain stimulation (transcranial direct current stimulation; tDCS) to reduce reactivity to personal urgency cues and attenuate symptoms of UUI. This is a novel step towards providing personalized efficacious non-pharmacologic treatment for UUI.

DETAILED DESCRIPTION:
Urinary urgency incontinence (UUI) is a highly prevalent, morbid and costly (up to $83 billion/year) disorder among older women, with up to 36% of those over 65 afflicted. One commonly experienced phenomenon among those with UUI is conditioned bladder responses to external triggers, often labeled "situational incontinence." Situational incontinence is described by sufferers as urinary urgency and leakage when confronted with specific contextual triggers or cues, such as approaching the front/garage door 'latch-key incontinence', and exposure to running water such as doing dishes. Generally ascribed to 'bladder spasms' (detrusor overactivity), studies have revealed that anywhere between 42% and 80% of women with UUI experience situationally provoked urgency, with approximately 26% of those experiencing situationally triggered leakage. The researchers recent work has focused on developing methods to recreate exposure to individuals' situational urgency cues, testing the impact of "urgency" and "safe" cues on self-report urgency and actual leakage, and finally assessing the role of bladder control mechanisms in the brain in response to these personal situational cues. The researchers found that women with situational UUI experienced increased urgency and leakage when exposed to personal "urgency" versus "safe" photographic cues from their daily lives. Further, brain areas related to attentional and visuospatial processing were activated during exposure to urge, but not safe, cues. Past studies of urgency simulated by bladder filling, show that prefrontal cortex, a seat of executive control, is activated to aid in controlling bladder activation. However, the study found that the prefrontal cortex (PFC) was not recruited during exposure to visual cues among women with situational urgency. Thus, the researchers propose that interventions capable of enhancing PFC activation during exposure to urgency situations should enable women to gain executive control over cues and result in less cue-provoked urgency and leakage, as well as overall UUI symptomatology. Using these now well-tested methods to personalize stimuli with photographs of urgency-provoking situational cues, the goal is to test the feasibility, acceptability, and compliance of these promising methods to attenuate urgency-related reactivity and reduce UUI symptoms. These novel methods include: (1) Brief mindfulness (MI) focused on body scan and acceptance language, (2) Transcranial direct current stimulation (tDCS) applied to the dorsolateral PFC, and (3) a combination of MI + tDCS. Sixty women with situational UUI will be randomized into a 7-session study, with a mail-in follow up 1-week post-training. All participants will undergo 4 urgency-cue exposure training sessions during which they will engage in one of the three interventions, based on group. Changes in urgency will be assessed via pre-post training differences in: Cue-reactivity to personal urge and safe cues, reaction time to a urinary Stroop task, self-report severity of bladder problems, and UUI episodes and urgency ratings on a daily bladder diary. Attenuating reactivity to situational urgency cues will increase our ability to complement and enhance the efficacy of UUI therapy and reduce symptom burden for its many sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Female; 40+ years old
* Self-report situational urgency in at least 4 of 15 common scenarios
* At least 2 leaks/week
* Urge Urinary Incontinence symptomatology bother score ≥4

Exclusion Criteria:

* Cognitive impairment (inability to complete tasks) as measured by Montreal Cognitive Assessment (MoCA) score < 26
* Urinary retention (PVR>200ml)
* Interstitial cystitis
* Spinal cord injury
* Pelvic irradiation or other cause of pelvic nerve damage
* Active urinary tract infection (UTI)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Conklin, PhD, Principal Investigator — University of Pittsburgh; Becky Clarkson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication, no end date
Access Criteria: Any purpose

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred by telephone screening respondents to research registries (Pitt+Me and the Pepper Research Registry of Older Adults), online advertising, other advertisements (flyers in senior centers and public places i.e. libraries, coffee shops, senior centers, hospital noticeboards), and referrals from the Benedum Geriatric center, local urogynecologists and urologists, faculty geriatricians, and local women's health and continence centers.
Pre-assignment Details: Participant exclusion prior to randomization occurred if the participant did not have enough urgency places, failed a urine screen, did not react to urgency cues at pre-test cue-reactivity, or chose not to continue participation after session 1.
Period: Overall Study
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Started (Started intervention) | 20 | 21 | 20
Completed | 20 | 19 | 20
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS | Total
Number analyzed (Participants) | 20 | 21 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 9 | 40
  >=65 years | 6 | 4 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.8) | 58.0 (8.9) | 64.8 (12.8) | 60.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 20 | 61
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 19 | 20 | 19 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 14 | 15 | 16 | 45
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Procedures Measured by Percentage of Participants Starting Intervention Who Complete the Study
Description: Feasibility is measured as the number of participants who completed the study divided by the total number of participants who started the intervention.
Time Frame: 4-weeks post intervention
Population: Number of participants that started the intervention (i.e. attended the first intervention visit) was 61. Thus, 61 participants started the intervention, and 59 participant completed all visits and intervention procedures
Measure: Number; unit: percentage of participants who completed
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 20 | 21 | 20
percentage of participants who completed | 100 | 90.4 | 100

2. Primary Outcome: Acceptability of Study Procedures
Description: Acceptability of study procedures was measured by 8-items assessing burden, difficulty, likeability of the study procedures on a 0-100 scale on the Post-Study Survey. A higher score indicates greater acceptability.
Time Frame: 4-weeks post intervention
Population: Analysis is based on number of mail-in acceptability questionnaires returned. Questionnaires were not returned for 2 participants in the transcranial direct current stimulation(tDCS) group and 2 participants in the Mindfulness group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 18 | 17 | 20
score on a scale | 85.6 (9.9) | 83.4 (13.6) | 80.4 (12.8)

3. Primary Outcome: Compliance With Study Procedures
Description: Compliance with study procedures measured by 2-items with a 0-100 scale on the Post-Study Survey. A higher score indicates greater compliance.
Time Frame: 4-weeks post intervention
Population: Transcranial Direct Current Stimulation group did not answer mindfulness compliance question. Analysis is based on number of mail-in acceptability questionnaires returned. Questionnaires were not returned for 2 participants in the transcranial direct current stimulation(tDCS) group and 2 participants in the Mindfulness group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 18 | 17 | 20
score on a scale
  Diary Compliance | 88.3 (12.9) | 84.1 (9.4) | 90.5 (10.0)
  Mindfulness Compliance: number analyzed (Participants) | 18 | 0 | 20
  Mindfulness Compliance | 94.4 (8.6) |  | 93.0 (10.3)

4. Primary Outcome: Change From Baseline to Post-intervention in Cue-induced Reactivity to Personal Photographic Urge Cues.
Description: Urinary urgency in response to personal photographic cues was self-reported by participants on 4 post-picture trial questions. Ratings were done using a 0-100 scale. The 4 items were averaged to calculate an urgency cue rating and safe cue rating for each picture trial. An overall Cue reactivity urgency rating was calculated for each participant by averaging their total urgency cue trial ratings. The same was done for safe cues.
  Cue reactivity was calculated as the difference between the overall rating averages for urgency cues and safe cues.
  Cue reactivity post-intervention was subtracted from that calculated for baseline. A lower score indicates greater reduction in cue-reactivity
Time Frame: Baseline (pre-intervention) to 1 week after completion of intervention activities
Population: Due to computer error at the time of data collection, data were not collected for three participants for this analysis (one per group).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 19 | 18 | 19
score on a scale | -25 (20) | -35 (13) | -19 (18)

5. Primary Outcome: Reaction Time to Urinary Stroop Task
Description: Change in reaction time to words associated with urgency from baseline to post-intervention. A lower score indicates greater reduction in reaction time.
Time Frame: Baseline (pre-intervention) to 1 week after completion of intervention activities
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 19 | 18 | 19
milliseconds | -36.95 (102.25) | -16.89 (87.30) | -81.63 (78.31)

6. Primary Outcome: Change From Baseline in Severity of Bladder Problem Measured by the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS)
Description: Change from baseline in severity of bladder problem measured by the ICIQ-FLUTS (International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms) a 12-item questionnaire (each item rated 0-4) evaluating urinary tract symptoms and impact on quality of life. A higher total score indicates greater symptoms and greater impact on quality of life. Score range (0-48) ICIQ-FLUTS was completed at baseline (pre-intervention) and one week after completion of all intervention activities. Pre-intervention score was subtracted from post-intervention score. A more negative score indicates greater symptom reduction.
Time Frame: Baseline (pre-intervention) to 1 week after completion of intervention activities
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 20 | 19 | 20
score on a scale | -2.65 (0.79) | -2.36 (0.81) | -2.10 (0.79)

7. Primary Outcome: Change in Number of Urge Urinary Incontinence (UUI) Episodes After Intervention
Description: Change in the number of Urge Urinary Incontinence (UUI) episodes was calculated from the mean number of incontinence episodes per day reported on a 3-day bladder diary pre-treatment and mean the number of UUI episodes per day on a 7-day bladder diary measured the week immediately after intervention concluded (post treatment). Post-intervention mean was subtracted from baseline mean. A more negative score indicates greater reduction in UUI episodes.
Time Frame: Baseline (pre-intervention) to 1 week after completion of intervention activities
Measure: Mean (Standard Error); unit: Number of incontinence episodes/day
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
Number analyzed (Participants) | 20 | 19 | 20
Number of incontinence episodes/day | -0.81 (0.23) | -0.90 (0.24) | -0.95 (0.23)

ADVERSE EVENTS:
Time Frame: 1 year 6 months (entire recruitment period)
Arm/Group | Mindfulness Training | Transcranial Direct Current Stimulation (tDCS) | Mindfulness + tDCS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04652869/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04652869/SAP_001.pdf